CLINICAL TRIAL: NCT05596994
Title: Use of 7T Multimodal Imaging to Detect Brain Changes Associated With Light Therapy in Persons With Mild Cognitive Impairment and Mild Alzheimer's Disease
Brief Title: 7T MRI for Light Therapy in Patients With Mild Cognitive Impairment and Mild AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Priti Balchandani, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 21-0668; R21AG076211 (NIH)
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light Intervention Therapy (LIT) then Sham LIT (Active Comparator): The LIT will begin at the patient's home and will be presented for 10 weeks. A washout period of 1 month will be scheduled to diminish carryover effects of the first therapy arm, then patients will begin the Sham LIT.
  Interventions: Device: Lighting Intervention Therapy; Device: Sham LIT
- Sham LIT then Light Intervention Therapy (Active Comparator): LIT will be performed identical to Arm 1, except for switchover of active LIT and Sham. A washout period of 1 month will be scheduled to diminish carryover effects of the LIT arm.
  Interventions: Device: Lighting Intervention Therapy; Device: Sham LIT

INTERVENTIONS:
Device: Lighting Intervention Therapy — The LIT will provide high circadian stimulation during the day produced by light sources that provide moderate light levels of spectra that are tuned to the sensitivity of the circadian system. The TLI intervention will remain in place and will be delivered to participants for 10 weeks each in a counterbalanced manner. Combining spectrum and light level, LIT will allow the research team to: (a) use a light source that will stimulate the circadian system, and (b) provide the participants with options as to how the light treatment will be delivered. The research team will deliver at least 300-400 lux at the eye of the bluish-white light during the day (CS of 0.4 or greater) and about 50 lux at the eye during the evening hours (CS of less than 0.1) and when the control lighting intervention is used.
Device: Sham LIT — A placebo comparison lighting intervention will be used. The comparison lighting intervention will remain in place and will be delivered to participants for 10 weeks.

SUMMARY:
The purpose of this research study is to investigate the effect of a light treatment on sleep, memory and brain function. In people with mild cognitive impairment (MCI) and Alzheimer's disease, sleep-wake disturbance is evident in up to 60% of patients. This can be caused by disruption of circadian rhythms and may affect our health and well-being. Circadian rhythms are the natural cycle of physical, mental, and behavior changes that the body goes through in a 24-hour cycle. Circadian rhythms are mostly affected by light and darkness and are controlled by a small area in the middle of the brain. They can affect sleep, body temperature, hormones, appetite, and other body functions. The circadian system plays an important role in the body and can affect sleep and brain function.

The results of the research would help develop light-delivery methods to improve sleep and memory in patients with mild cognitive impairment (MCI) and Alzheimer's disease who typically spend a significant amount of time indoors.

DETAILED DESCRIPTION:
Subjects will be enrolled in the study for 26 weeks. During the first week, subject will come in to Mount Sinai for a study visit to complete a few questionnaires about sleep and mood, complete several memory tests and have an MRI of their brain. These study visits will take about 2 hours to complete. During this week, subject will also be asked to wear a wrist actigraph and light meter for 7 days. The actigraph is similar in size to a watch and is used to record their activity and rest patterns, and the light meter measures the amount of light they are exposed to during the day. After the completion of this week, subject will have a light treatment installed in their home that will be in place for 10 weeks. During the last week of the light treatment, subject will again come into Mount Sinai and repeat the questionnaires, memory tests and MRI, and wear the actigraph and light meter. After a 4-week break, subject will again come into Mount Sinai for a third study visit and complete the same questionnaires, memory tests, and MRI, and wear the actigraph and light meter. After this week, subject will have a different type of light treatment installed in their home and left in place for 10 weeks. During the last week of the light treatment, subject will come into Mount Sinai for the final study visit and complete the questionnaires, memory tests and MRI, and wear the actigraph and light meter for 7 days. There are no costs associated with participation, but subject will receive monetary compensation for each of the 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* the patients must have undergone PET scans to measure amyloid protein accumulation within the past year
* Those taking antidepressants will be included, but type of medicine and dosage intake will be monitored.
* 50 years and older
* Eligible participants will be amnestic mild cognitive impairment (MCI) or mild Alzheimer's disease (AD) patients with circadian sleep disturbances who reside in their homes, independent living, or assisted living facilities.
* confirmed amyloid beta positive from an existing ADRC cohort with PET scan (age: 50-85 yrs, 40% M, 60% F; falling between 0.5-4.0 and 4.5-9.0 in the Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB)

Exclusion Criteria:

* Those taking sleep medication will be not included
* Presence of another brain disease that fully explains the dementia (extensive brain vascular disease, Parkinson's disease, dementia with Lewy bodies, traumatic brain injury, or multiple sclerosis)
* residence in a skilled nursing facility or long-term care
* indication for psychiatric hospitalization or acute suicidality in the opinion of the physician
* recent changes in psychotropics (14 days)
* major organ failure (e.g., kidney failure)
* uncontrolled generalized disorders such as hypertension or diabetes
* obstructing cataracts, macular degeneration, and blindness

  o Those who have undergone cataract surgery and received an intraocular lens coated with ultraviolet- and blue-blocking filters (400-440/440-500 nm) will also be excluded
* severe sleep apnea:

  o Apnea will be screened for using the Sleep Apnea scale of the Sleep Disorders Questionnaire (SA-SDQ), a 12-item scale yielding scores between 0 and 60.3. The study will use a score of 29 as a cutoff for men (sensitivity 75%, specificity 65% for sleep apnea), and a cutoff of 26 for women (sensitivity 80%, specificity 67%).
* restless leg syndrome (RLS):

  o RLS will be screened for using the International Restless Legs Scale (IRLS), a 10-item scale that yields scores between 0 and 40.4 The study will use a cutoff of greater than or equal to 11 (indicating the presence of symptoms that are at least moderate) as a positive screen for RLS
* history of:

  * severe photosensitivity dermatitis
  * severe progressive retinal disease (e.g., macular degeneration), or;
  * a permanently dilated pupil (e.g., after certain types of cataract surgery)
* 7T MRI specific exclusions including presence of metallic or biomedical implants (patients can be enrolled at the discretion of the study team and site MRI technicians) and claustrophobia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in Brian Volumes | Baseline and post-therapy at Week 26
  Volumes of structures associated with cognitive impairment and AD pathophysiology will be quantified from 7T imaging data. Hippocampal subfield volumes and amygdala subnuclei volumes will be computed. The measures will be compared pre- and post-therapy to determine effect of LIT on the brain.
Changes in Perivascular Space Density | Baseline and post-therapy at Week 26
  Perivascular spaces will be computed from structural scans using automated segmentation methods. The measures will be compared pre- and post-therapy to determine effect of LIT on the brain.

SECONDARY OUTCOMES:
Changes in Structural connectivity as measured by dMRI | Baseline and post-therapy at Week 26
  Diffusion magnetic resonance imaging (dMRI) will be performed. DMRI quantifies the freedom of water molecules to diffuse in various directions, providing information on the microstructural properties of tissues, including diffusivities, fractional anisotropy (FA, the degree to which diffusivity differs with respect to direction, which indicates structural integrity of axons), and the vector along which diffusion is least restricted (which corresponds to the direction of nerve axons in the brain). From these measures, probabilistic streamlines are generated between various brain regions. The number of streamlines connecting two brain regions gives an indication of the degree to which they are connected by axons. Various network theory measures can be generated for each brain region based on a mathematical analysis of its structural connections to other regions. The measures will be compared pre- and post-therapy to determine effect of LIT in the structural connectivity.
Changes in Functional connectivity as measured by fMRI | Baseline and post-therapy at Week 26
  Functional magnetic resonance imaging (fMRI) will be performed. FMRI is sensitive to the amount of deoxygenated blood in a given region of the brain, which varies in response to changes in nerve activation in that region, and in an fMRI experiment, a time series of images is taken over the course of several minutes such that a time-course of neural activation is recorded at each location in the brain In resting-state fMRI, the degree to which the time-course of neural activation in a region of the brain is correlated to the time-course of neural activation in another region of the brain is taken as an indication of the degree to which they are functionally connected. Various network theory measures can be generated for each brain region based on a mathematical analysis of its functional connectivity to other regions. The measures will be compared pre- and post-therapy to determine effect of LIT in the functional connectivity.
Percentage of Time Spent in Bed Sleeping | 7 days/week for 26 weeks
  Sleep efficiency will be calculated as the percentage of time spent in bed sleeping using Actigraphy.
Pittsburgh Sleep Quality Index (PSQI) Score | Baseline and every 4 weeks for duration of the study
  Sleep disturbance using The Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-rated 19-item questionnaire which assesses sleep quality and disturbances. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall global score ranging from 0 to 21, where lower scores denote a healthier sleep quality, higher score indicates worse sleep quality. A global score >5 is considered to indicate sleep disturbance.
Circadian Stimulus (CS) values using the Daysimeter | During waking hours for 26 weeks
  Light exposure will be measured by the Daysimeter. The instrument will measure photopic light levels (lux) and circadian light levels received by the subject during the day when they are wearing the pendant/pin. This data will then be used to calculate the circadian stimulus (CS) values the subjects are receiving.
Changes in Montreal Cognitive Assessment (MoCA) Score | Baseline and at the end of each intervention period (each intervention period is 10 weeks)
  Changes in cognitive status using the Montreal Cognitive Assessment (MoCA). The MoCA is a 1-page, 30-point test that can be administered in 10 minutes. It assesses short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. In a validation study, it was shown to be a promising tool for detecting mild cognitive impairment and early Alzheimer's onset compared to the MMSE. Total scores for MoCA range from 0-30, where higher scores indicate better health outcomes.
Changes Geriatric Depression Scale (GDS) Score | Baseline and at the end of each intervention period (each intervention period is 10 weeks)
  Changes in depression using the GDC Score. The GDS is an instrument used to measure depression in healthy adults. This study will use a short version of the GDS consisting of 15 questions. Ten of the questions indicate the presence of depression when answered positively, and the other five questions indicate depression when answered negatively. Scores of 0-4 = normal, 5-8 = mild depression, 9-11 = moderate depression, and 12-15 = severe depression. Total scale ranges from 0-15, where higher scores indicate more severe depression.
Changes in Dementia Quality of Life Instrument (DQoL) Score | Baseline and at the end of each intervention period (each intervention period is 10 weeks)
  Changes in Quality of Life using the DQoL. The DQoL is designed to assess health-related QoL in persons suffering from dementia. It is administered in interview format, with information obtained exclusively from the elder. The DQoL measures self-esteem, positive affect/humor, negative affect, feelings of belonging, and sense of aesthetics. The DQoL consists of 29 items, grouped into 5 subscales according to domain. Each of the subscales have a possible range of 1-5, where a higher score indicates better QoL. The subscale scores are not summed for an overall measure of QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Priti Balchandani, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot exploratory study.